CLINICAL TRIAL: NCT05506761
Title: Ultrasound-Guided Continuous Rhomboid Intercostal Block Combined With Sub-Serratus Plane Block Versus Continuous Erector Spinae Plane Block for Analgesia in Patients With Multiple Traumatic Rib Fractures
Brief Title: Rhomboid Intercostal Block Combined With Sub-Serratus Plane Block Versus Erector Spinae Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Mahmoud ElNawagy, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 35167/12/21
Record Dates: First submitted 2022-08-17; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Rib Fractures
Keywords: Rib Fractures; Intercostal nerve block
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (No Intervention): This group includes patients with rib fractures receiving patient-controlled analgesia.
- Group II (Experimental): This group includes patients with rib fractures receiving continuous ultrasound-guided erector spinae plane block.
  Interventions: Procedure: ultrasound-guided erector spinae plane block
- Group III (Experimental): This group includes patients with rib fractures receiving continuous ultrasound-guided rhomboid intercostal block combined with sub-serratus plane block.
  Interventions: Procedure: ultrasound-guided rhomboid intercostal block combined with sub-serratus plane block

INTERVENTIONS:
Procedure: ultrasound-guided erector spinae plane block — Patients will receive 20 ml plain bupivacaine 0.25 % bolus, then 10 ml per hour plain bupivacaine 0.125 % continuous infusion via ultrasound-guided erector spinae plane block
  Arms: Group II
Procedure: ultrasound-guided rhomboid intercostal block combined with sub-serratus plane block — Patients will receive 20 ml plain bupivacaine 0.25 % bolus, then 10 ml per hour plain bupivacaine 0.125 % continuous infusion via ultrasound-guided rhomboid intercostal block combined with sub-serratus plane block
  Arms: Group III

SUMMARY:
The aim of this study is to assess the quality of analgesic efficacy and improvement of pulmonary function in patients with fracture ribs receiving either continuous rhomboid intercostal block combined with sub-serratus block or continuous erector spinae plane block by comparing and evaluating the differences between the two techniques.

DETAILED DESCRIPTION:
Rib fractures are common injuries usually following blunt thoracic trauma. Depending on the extent of the injury, rib fractures are associated with a high risk of pulmonary complications, requirement for critical care admission and mechanical ventilation with increased risk of mortality, especially in older patients.

Thoracic pain caused by rib fractures or chest contusion limits patients' coughing and deep breathing, which may cause atelectasis and pneumonia. Patients may also suffer from pulmonary contusion due to injuries and this situation may cause acute respiratory distress syndrome and/or respiratory failure.

The key points in the management of patients with rib fractures are a combination of adequate pain control, respiratory support and physiotherapy.

Previously, pain control of rib fractures has been managed with systemic analgesia alone, with only a minority of patients receiving regional anesthesia. The presence of comorbid conditions, debility and alterations in pharmacodynamics/pharmacokinetics in older patients often results in a higher incidence of adverse effects with systemic analgesia, especially when opioid analgesia is required.

Therefore, different kinds of analgesic techniques have been proposed, including epidural analgesia, local anesthetic infiltration, erector spinae plane (ESP) block, paravertebral block and serratus plane block (SAB) or a combination of the mentioned methods are used to relieve pain.

Erector spinae plane block (ESB) is a novel myofascial plane block introduced into clinical practice. It has been successfully utilized in the management of pain after both rib fractures and surgery of the abdomen and thorax, and in the management of chronic thoracic pain.

The ultrasound-guided rhomboid intercostal block (RIB) and rhomboid intercostal block combined with the sub-serratus plane (RISS) block are two new analgesic techniques work by anesthetizing the lateral cutaneous branches of the thoracic intercostal nerves and can be used in multiple clinical settings for chest wall and upper abdominal analgesia.

This study suggests that the use of ultrasound-guided continuous ESPB or continuous RIB may improve the analgesia in patients with multiple fracture ribs, decrease the opioid analgesia consumption, and improve the outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 21 - 60 years.
* Patients with blunt chest trauma.
* Multiple fracture ribs (at least 3 ribs).
* Patients with acute trauma less than 48 hours.

Exclusion Criteria:

* Patients with major trauma outside the chest wall e.g., severe traumatic brain injury or major abdominal visceral injuries.
* Patients with bilateral rib fractures.
* Patients that are intubated and mechanically ventilated.
* Pregnant Individuals.
* Patients with local deformity or infection at the site of injection.
* Sensitivity to local anesthetic drugs.
* Patients with flail chest.
* Patients with Suspected or diagnosed coagulopathy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid analgesic consumption per day | 4 days

SECONDARY OUTCOMES:
change in pain scores by Numerical rating score (NRS) after the procedure | 4 days
Time to First rescue analgesic request. | 4 days
Patient satisfaction. | 4 days
Changes in heart rate. | 4 days
Changes in mean arterial blood pressure. | 4 days
Incidence of adverse effects. | 4 days
Incidence of respiratory complications. | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peek J, Beks RB, Hietbrink F, Heng M, De Jong MB, Beeres FJP, Leenen LPH, Groenwold RHH, Houwert RM. Complications and outcome after rib fracture fixation: A systematic review. J Trauma Acute Care Surg. 2020 Aug;89(2):411-418. doi: 10.1097/TA.0000000000002716. PMID 32282759
- [Background] Bachoumas K, Levrat A, Le Thuaut A, Rouleau S, Groyer S, Dupont H, Rooze P, Eisenmann N, Trampont T, Bohe J, Rieu B, Chakarian JC, Godard A, Frederici L, Gelinotte S, Joret A, Roques P, Painvin B, Leroy C, Benedit M, Dopeux L, Soum E, Botoc V, Fartoukh M, Hausermann MH, Kamel T, Morin J, De Varax R, Plantefeve G, Herbland A, Jabaudon M, Duburcq T, Simon C, Chabanne R, Schneider F, Ganster F, Bruel C, Laggoune AS, Bregeaud D, Souweine B, Reignier J, Lascarrou JB. Epidural analgesia in ICU chest trauma patients with fractured ribs: retrospective study of pain control and intubation requirements. Ann Intensive Care. 2020 Aug 27;10(1):116. doi: 10.1186/s13613-020-00733-0. PMID 32852675
- [Background] Ostermann RC, Joestl J, Lang N, Tiefenboeck TM, Ohnesorg S, Platzer P, Hofbauer M. Thoracic Injuries in Pediatric Polytraumatized Patients: Epidemiology, Treatment and Outcome. Injury. 2021 Jun;52(6):1316-1320. doi: 10.1016/j.injury.2021.02.033. Epub 2021 Feb 17. PMID 33663803
- [Background] Dogrul BN, Kiliccalan I, Asci ES, Peker SC. Blunt trauma related chest wall and pulmonary injuries: An overview. Chin J Traumatol. 2020 Jun;23(3):125-138. doi: 10.1016/j.cjtee.2020.04.003. Epub 2020 Apr 20. PMID 32417043
- [Background] Warfield DJ Jr, Barre S, Adhikary SD. Current understanding of the fascial plane blocks for analgesia of the chest wall: techniques and indications update for 2020. Curr Opin Anaesthesiol. 2020 Oct;33(5):692-697. doi: 10.1097/ACO.0000000000000909. PMID 32826623
- [Background] O'Connell KM, Patel KV, Powelson E, Robinson BRH, Boyle K, Peschman J, Blocher-Smith EC, Jacobson L, Leavitt J, McCrum ML, Ballou J, Brasel KJ, Judge J, Greenberg S, Mukherjee K, Qiu Q, Vavilala MS, Rivara F, Arbabi S. Use of regional analgesia and risk of delirium in older adults with multiple rib fractures: An Eastern Association for the Surgery of Trauma multicenter study. J Trauma Acute Care Surg. 2021 Aug 1;91(2):265-271. doi: 10.1097/TA.0000000000003258. PMID 33938510
- [Background] Jiang CW, Liu F, Zhou Q, Deng W. Comparison of rhomboid intercostal nerve block, erector spinae plane block and serratus plane block on analgesia for modified radical mastectomy: A prospective randomised controlled trial. Int J Clin Pract. 2021 Oct;75(10):e14539. doi: 10.1111/ijcp.14539. Epub 2021 Jul 2. PMID 34133831
- [Background] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545